CLINICAL TRIAL: NCT04847011
Title: Deciphering the Impact of Exposures From the Gut Microbiome-derived Molecular Complex in Human Health and Disease
Acronym: ExpoBiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andreas Michalsen (Other)
Collaborators: University of Luxembourg (Other); Paracelsus Elena Klinik (Other)
Responsible Party: Sponsor-Investigator, Andreas Michalsen, Prof. Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ExpoBiome
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis; Parkinson Disease; Healthy
MeSH Terms: conditions — Arthritis, Rheumatoid; Parkinson Disease | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- RA - longitudinal arm (Experimental)
  Interventions: Other: Fasting
- PD - longitudinal arm (Experimental)
  Interventions: Other: Fasting
- RA - crosssectional arm (No Intervention)
- PD - crossectional arm (No Intervention)
- Healthy controls - crosssectional arm (No Intervention)

INTERVENTIONS:
Other: Fasting — Patients undergo a 5-10 day fasting period with a dietary energy supply 350-400kcal per day with fruit and vegetable juices or, if not feasible, an established fasting-mimicking diet of 600-800 kcal according to Longo et al.
  Arms: PD - longitudinal arm; RA - longitudinal arm

SUMMARY:
The ExpoBiome project will analyze the impact of fasting on patients with Parkinsons's Disease (PD) or rheumatoid arthritis (RA) on a clinical level as well as the effect of fasting on their immune system and gut microbiota. ExpoBiome will combine metagenomics and other "omics" [meta-transcriptomics, meta-proteomics and (meta-)metabolomics], bioinformatic analyses and biostatistics under a systems biology framework to gain new mechanistic insights into microbiome-immune system interactions in the context of chronic diseases with inflammatory signatures.

Besides a one time crossectional study of healthy participants, patients with RA and PD a longitudinal fasting study with two arms (RA and PD) is planned.

DETAILED DESCRIPTION:
The human gut microbiome is a complex ecosystem, which contributes essential functions to human physiology. Changes to the microbiome are associated with several chronic diseases characterised by inflammation, including neurodegenerative and autoimmune diseases. Microbiome-derived effector molecules comprising nucleic acids, (poly)peptides and metabolites are present at high levels in the gut but have so far eluded systematic study. This gap in knowledge is limiting mechanistic understanding of the microbiome's functional impact on chronic diseases such as Parkinson's Disease (PD) and rheumatoid arthritis (RA). Here, for the first time a combination of advanced high-resolution methodologies will be integrated to comprehensively identify the constituents of this molecular complex and their impact on the human immune system. First, a quantitative, integrated multi-omic analysis on microbiome samples collected from healthy individuals and patients with newly diagnosed PD or RA will be performes.

Using contextualised prior knowledge (ExpoBiome Map) and machine learning methods, we will identify microbial molecules associated with condition-specific immunophenotypes. Second, the biomarker signature during a model clinical intervention (therapeutic fasting) will be validated and tracked to predict treatment outcomes. Third, microbes and molecules will be screened in personalised HuMiX gut-on-chip models to identify novel anti-inflammatory compounds. By providing mechanistic insights into the molecular basis of human-microbiome interactions, the project will generate essential new knowledge about causal relationships between the gut microbiome and the immune system in health and disease. By facilitating the elucidation of currently unknown microbiome-derived molecules, it will identify new genes, proteins,metabolites and host pathways for the development of future diagnostic and therapeutic applications.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses: rheumatoid arthritis (first diagnosis >6 weeks ago and <8 years), parkinson's disease OR healthy volunteer
* Control ("healthy") individuals must be without any evidence of active, known or treated RA, without any evidence of active, known or treated central nervous system disease, and without a known family history of idiopathic PD
* Arthritis in at least one joint
* Control individuals should match the RA or PD individuals as closely as possible, especially their age, sex, and education
* Present written declaration of consent
* Consent to specimen collection and specimen use
* Ability to understand the patient information and willingness to sign the consent form

Exclusion Criteria:

* gout or proven bacterial arthritis
* Psychiatric illness that limits understanding of the examination protocol (unable to consent)
* BMI < 18.5
* Pre-existing/current eating disorders (bulimia nervosa, anorexia nervosa) within the past 5 years.
* Severe internal diseases (e.g. renal insufficiency with creatinine > 2mg/dl)
* Participation in another study
* Existing vegan diet or fasting within the past 6 months
* Pregnancy or breastfeeding
* Chronic inflammatory bowel disease
* Use of antibiotics within the past 12 months
* Presence of anemia

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Gut microbiota Characterization | Change over baseline to 12 months
  Molecular typing of the gut microbiota using sequencing and high-throughput analysis from stool samples (metagenomics, metatranscriptomics, metaproteomics, metabolomics)

SECONDARY OUTCOMES:
Resting blood pressure | Change over baseline to 12 months
Heart rate | Change over baseline to 12 months
Abdominal circumference | Change over baseline to 12 months
Waist to Hip Ratio | Change over baseline to 12 months
Body Mass Index (kg/m2) | Change over baseline to 12 months
Disease Activity Score 28 (DAS-28-CRP) | Change over baseline to 12 months
  Change from Baseline in the DAS-28-CRP, range from 2.0 to 10.0 while higher values meaning a higher disease activity and below of 2.6 meaning remission
Health Assessement Questionnaire (HAQ) | Change over baseline to 12 months
  Change from Baseline in the HAQ, range from 0 to 3 while higher values meaning a higher grade of disability
Simplified Disease Activity Index Score (SDAI) | Change over baseline to 12 months
  Change from Baseline in the SDAI, range from 0 to 86 with assumed range from 0.1 to 10mg/dL for CRP. Higher values mean a higher disease activity and below of 34 meaning remission.
Hannover Functional Ability Questionnaire (Funktionsfragebogen Hannover, FFbH-R) | Change over baseline to 12 months
  Change from Baseline in the FFbH-R, range from 0 to 100 % while higher values meaning a higher grade of functional capacity
MDS-UPDRS | Change over baseline to 12 months
  Movement Disorders Society-sponsored revision of the Unified Parkinson's Disease Rating Scale part I, II, IV (MDS-UPDRS part I, II, IV). Total score range: 0-260 (including the MDS-UPDRS part III), including 4 subcategories. Subcategories are summed to compute the total score. A lower score means a better outcome.
Parkinson's Disease Sleep Scale-2 (PDSS-2) | Change over baseline to 12 months
  The Parkinson's Disease Sleep Scale 2 (PDSS-2) is designed to assess nocturnal disability in Parkinson's disease. The PDSS-2 is a 15 question analog scale that ranks answers from 0 - 4, with 4 being worse. (Question 1 is an exception, where 4 is better and 0 is worse). In addition to an overall assessment of sleep disability three aspects of sleep problems can be obtained; disturbed sleep (total of questions 1-3, 8 and 14), PD-specific nocturnal motor symptoms (total of questions 4-6, 12 and 13), and PD-specific nocturnal symptoms (Total of questions 7, 9-11 and 15).
Parkinson's Disease Questionnaire-39 (PDQ-39) | Change over baseline to 12 months
  The 39 question Parkinson's Disease Questionnaire (PDQ-39) is a patient-reported rating scale for quality of life in Parkinson's disease. Respondents affirm if they have experienced problems due to their disease using a five point scale from never (0 points) to always (4 points, or worse) in doing common activities. The PDQ-39 is comprised of 8 domains: mobility, emotion, activities of daily living, cognition, stigma, social support, communication, bodily discomfort. Total possible range of scores = 0 - 156, with higher scores representing worse severity.
Non-motor symptoms questionnaire (NMSQ) | Change over baseline to 12 months
  The non-motor symptoms (NMS) questionnaire can be given to people affected by Parkinson's in order to aid health and social care professionals to assess their non-motor symptoms.The non-motor symptoms questionnaire is a 30-point, patient-based questionnaire used to determine the non-motor symptoms experienced by the patient during the past month. The points should be totalled to give a score out of 30. A score of under 10 is mild, 10-20 moderate and over 20, severe.
Non Motor Symptoms Scale (NMSS) | Change over baseline to 12 months
  The Non-Motor Symptoms Scale (NMSS) measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease, through 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe). Frequency is rated on a scale from 1 (rarely) to 4 (very frequent). Item scores are calculated as the product of severity and frequency; the total score is obtained by summing the item scores. The NMSS total score ranges from 0 to 360 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms (reduced score).
Stress questionnaire (Cohen Perceived Stress Scale, CPSS) | Change over baseline to 12 months
  Change from Baseline in the CPSS, range from 0 to 4 in each item. Scores are obtained by reversing responses (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) to the positively stated items and then summing across all scale items, higher values meaning a higher grade of perceived stress.
Quality of Life questionnaire (WHO-5) | Change over baseline to 12 months
  Change from Baseline in the WHO-5, range from 0 to 100 %, higher values meaning a higher grade of well-being
Hospital Anxiety and Depression Scale (HADS) | Change over baseline to 12 months
  Assessing full scale, range 0-42, lower score meaning a better outcome
Mood questionnaire (Profile of Mood States, POMS) | Change over baseline to 12 months
  Change from Baseline in Emotional Distress will be measured using the German Version of the Profile of Mood States (ASTS) short version (19 items, 7-point Likert scale; 0=not at all, 6=extremely). Lower scores indicate more stable mood profiles.
Sociodemographic Measurements | Baseline
  Age, gender, education level, household income, employment status, marital status, language spoken, complete family history, current and previous illness and co-morbidities, and current medications
Behavioral Factors | Change over baseline to 12 months
  Physical inactivity, coffee, health promoting activities via Likert Scales, range from 0 to 5 while higher values meaning a higher grade of agreement
Dietary Behaviour | Change over baseline to 12 months
  Modified FFQ recording dietary behaviour such as mealtimes, frequency of food intake, food preferences, fasting experiences
Behavioral Factors: alcohol consumption | Change over baseline to 12 months
  Number of alcoholic beverages on average per week in the last month
Behavioral Factors: smoking | Baseline
  Smoking status in packyears
Expectation questions | Baseline
  For fasting on a 5-point likert scale from 1 (nothing at all) to 5 (very strong)
Differential blood count | Change over baseline to 12 months
Hepatic transaminases (GPT, GOT) and Gamma glutamyl transpeptidase (y-GT) | Change over baseline to 12 months
  GPT in units per liter (U/L) GOT (U/L) y-GT (U/L)
Bilirubine (total, direct, indirect in mg/dL) | Change over baseline to 12 months
Total protein in grams per liter (g/L) | Change over baseline to 12 months
Albumine in grams per liter (g/L) | Change over baseline to 12 months
Creatinine in µmol per liter (µmol/L) | Change over baseline to 12 months
Estimated glomerular filtration rate (eGFR) in milliliter per minute (mL/min) | Change over baseline to 12 months
Alcalic Phosphatase in units per liter (U/L) | Change over baseline to 12 months
Urea in milligrams per deciliter (mg/dL) | Change over baseline to 12 months
Blood lipids and fasting glucose | Change over baseline to 12 months
  * triglycerides (mmol/L)
  * total cholesterol (mmol/L)
  * LDL (mmol/L)
  * HDL (mmol/L)
  * fasting glucose (mmol/L)
HbA1C (mmol/mol Hb, %) | Change over baseline to 12 months
TSH (mU/L) | Change over baseline to 12 months
IGF-1 (ng/mL) | Change over baseline to 12 months
Insulin (mU/L) | Change over baseline to 12 months
High sensitive CrP (mg/L) | Change over baseline to 12 months
  Evaluate change in hs-CrP levels in participants with RA
Rheumatoid factor (RF, IgM) (U/mL) | Baseline
  Evaluate RF status in participants with RA
Anti-cyclic citrullinated peptide (ACPA) (U/mL) | Change over baseline to 12 months
  Evaluate change in ACPA levels in participants with RA
Zonulin (ng/mL) | Change over baseline to 12 months
Fatty acid binding protein 2 (FABP2) (pg/mL) | Change over baseline to 12 months
Plasma Calprotectin (µg/g) | Change over baseline to 12 months
Fecal Calprotectin (µg/g) | Change over baseline to 12 months
Phenotyping of immune cells | Change over baseline to 12 months
  Determination of cytometric parameters that indicate changes in cell activation or quantitative changes in the absolute and/or relative size of subpopulations (e.g. classical/intermediate/non-classical monocytes, naïve and memory T-cells, B-cell differentiation to plasmablasts/-cells) Gene expression analysis of immune cells with Affymetrix whole genome microarrays and RNAseq to search for transcriptional patterns and markers that help to identify relevant immune cell (sub-)populations, which are not yet included in the cytometric phenotyping screen
Urine metabolomics (10 ml midstream urine) | Change over baseline to 12 months
Oral microbiota analysis in saliva | Change over baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr. med., Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (2):
- Germany (2):
  - Paracelsus-Elena-Klinik Kassel, Kassel, Hesse
  - Charité Hochschulambulanz für Naturheilkunde am Immanuel Krankenhaus, Berlin

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Hansen B, Laczny CC, Aho VTE, Frachet-Bour A, Habier J, Ostaszewski M, Michalsen A, Hanslian E, Koppold DA, Hartmann AM, Steckhan N, Mollenhauer B, Schade S, Roomp K, Schneider JG, Wilmes P. Protocol for a multicentre cross-sectional, longitudinal ambulatory clinical trial in rheumatoid arthritis and Parkinson's disease patients analysing the relation between the gut microbiome, fasting and immune status in Germany (ExpoBiome). BMJ Open. 2023 Aug 18;13(8):e071380. doi: 10.1136/bmjopen-2022-071380. PMID 37597865